CLINICAL TRIAL: NCT04768634
Title: Predicting Arrhythmogenic Risk in Congenital Heart Patients: the PRECISION Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: limited enrollment
Sponsor: Boston Children's Hospital (Other)
Collaborators: American Heart Association (Other); The Children's Heart Foundation (Other)
Responsible Party: Principal Investigator, Audrey Dionne, Pediatric Cardiologist, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-P00037574
Record Dates: First submitted 2021-02-08; First posted 2021-02-24 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Arrhythmia in Children; Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observation (No Intervention): Patients will be observed for arrhythmias and treated if they occur.
- Testing (Experimental): Patients will undergo provocative electrophysiology testing, and antiarrhythmic medication considered if arrhythmias can be induced.
  Interventions: Diagnostic Test: Provocative electrophysiology study

INTERVENTIONS:
Diagnostic Test: Provocative electrophysiology study — Provocative electrophysiology testing will be performed at the bedside using the temporary pacing wires placed at the time of surgery.
  Arms: Testing

SUMMARY:
In this research study we want to learn more about abnormal heart rhythm after cardiac surgery in children. These abnormal heart rhythms, also called arrhythmias, may occur due to several reasons after cardiac surgery. They can be due to abnormal electrical pathway or an irritable area of the heart that stimulates abnormal impulses. Regardless of the cause, arrhythmias after cardiac surgery can be a problem, extending the hospital stay, requiring additional medications and even leading to cardiac arrest.

Current practice is to monitor for arrhythmias after cardiac surgery, and to treat them if they occur. With this research, we want to investigate whether we can identify patients who will develop arrhythmia, and treat them before they occur.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled trial of provocative electrophysiology testing and prophylactic treatment of inducible SVT versus expectant management

ELIGIBILITY:
Inclusion Criteria:

* Patients aged < 18 years of age on admission to the cardiac intensive care unit following cardiac surgery with a predicted probability of supraventricular tachycardia >10%

Exclusion Criteria:

* Patients following orthotopic heart transplant, ventricular assist device implantation, primary extracorporeal membrane oxygenation cannulation, pacemaker or implantable cardioverter-defibrillator implantation or sympathectomy
* Patients on antiarrhythmic medication at the time of surgery
* Patients with atrioventricular conduction disease (1st degree atrioventricular block with PR interval greater than 200 ms, 2nd degree atrioventricular block or complete heart block)
* Patients with severe ventricular dysfunction in whom therapy with beta-blocker or sotalol is deemed contra-indicated by the primary team
* Patients with absent or non-functioning atrial pacing wires

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Number of patients with supraventricular tachycardia | Through hospital discharge after cardiac surgery, or up to 90 days
  Number of days post-operatively at time of supraventricular tachycardia

SECONDARY OUTCOMES:
Number of patients with adverse events related to provocative electrophysiology testing | Through hospital discharge after cardiac surgery, or up to 90 days
Number of patients with sustained supraventricular tachycardia | Through hospital discharge after cardiac surgery, or up to 90 days
  Number of days post-operatively at time of sustained supraventricular tachycardia
Number of patients with other tachyarrhythmias | Through hospital discharge after cardiac surgery, or up to 90 days
Number of days post-operatively at time of extubation | Through hospital discharge after cardiac surgery, or up to 90 days
Number of days post-operatively in the intensive care unit | Though hospital discharge
Number of days in the hospital | Through hospital discharge after cardiac surgery, or up to 90 days
Number of patients with adverse events related to antiarrhythmic treatment | Through hospital discharge after cardiac surgery, or up to 90 days
Number of patients with major adverse cardiac events (including need for CPR, ECMO or death) | Through hospital discharge after cardiac surgery, or up to 90 days
Number of patients with supraventricular tachycardia after hospital discharge | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Dionne, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No